CLINICAL TRIAL: NCT00003619
Title: A Phase I/II Combination Study of Topotecan, Fludarabine, Cytosine Arabinoside and G-CSF (T-FLAG) Induction Therapy in Patients With Poor Prognosis AML, MDS and Relapsed/Refractory ALL Followed by Maintenance of Either PBSC Transplant or 13 Cis-Retinoic Acid
Brief Title: Combination Chemotherapy Followed By Peripheral Stem Cell Transplantation or Isotretinoin in Treating Patients With Acute Myeloid Leukemia, Myelodysplastic Syndrome, or Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: AUH-MCP-70612-01; CDR0000066698 (Registry Identifier: PDQ (Physician Data Query)); AUH-MCP-70612-02P; NCI-V98-1485
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2008-02

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Thrombocytopenia
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; polycythemia vera; primary myelofibrosis; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; chronic myelomonocytic leukemia; secondary acute myeloid leukemia; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; thrombocytopenia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Thrombocytopenia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Filgrastim; Vitamin E; Busulfan; Cytarabine; Etoposide; fludarabine phosphate; Isotretinoin; Topotecan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Dietary Supplement: vitamin E
Drug: busulfan
Drug: cytarabine
Drug: etoposide
Drug: fludarabine phosphate
Drug: isotretinoin
Drug: topotecan hydrochloride
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Isotretinoin may help cancer cells develop into normal white blood cells.

PURPOSE: Phase I/II trial of topotecan, fludarabine, cytarabine, and filgrastim followed by peripheral stem cell transplantation or isotretinoin in treating patients who have acute myeloid leukemia, myelodysplastic syndrome, or recurrent or refractory acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of topotecan in combination with fludarabine, cytarabine, and filgrastim (FLAG) in patients with poor prognosis acute myeloid leukemia, myelodysplastic syndrome, or recurrent or refractory acute lymphocytic leukemia. II. Determine the maximum tolerated dose of topotecan in the FLAG regimen in these patients. III. Assess the complete remission rates in patients treated with this regimen.

OUTLINE: Patients with complete response proceed to further therapy according to age. 65 and under: Patients receive etoposide by IV continuously for 5 days, cytarabine IV over 2 hours every 12 hours for 4 days, and filgrastim (G-CSF) subcutaneously. Peripheral blood stem cells (PBSC) are then harvested. Patients then receive oral busulfan every 6 hours on days -7 to -4 and etoposide IV over 10 hours on day -3. PBSC are reinfused on day 0. Over 65: Patients receive oral isotretinoin and vitamin E daily. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed every month for 1 year and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven poor prognosis acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or recurrent/refractory acute lymphocytic leukemia, including: Myelodysplastic syndrome (MDS) stages B and C Refractory anemia, refractory anemia with ringed sideroblasts, or refractory anemia with excess blasts (between 5% and 20% myeloblasts) MDS with increased erythroblasts or monocytoblasts of no greater than 20% MDS in transformation (between 20% to 30% myeloblasts) or acute nonlymphoblastic leukemia (at least 30% myeloblasts) Chronic myelomonocytic leukemia Poor prognosis refractory or recurrent acute myeloid leukemia after complete response Secondary or therapy related AML or MDS AML blastic crisis of chronic myelogenous leukemia or other myeloproliferative disorders such as polycythemia vera, essential thrombocytopenia, or agnogenic myeloid metaplasia

PATIENT CHARACTERISTICS: Age: 19 to 90 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT or SGPT less than 2.0 times upper limit of normal Renal: Normal serum creatinine Cardiovascular: No congestive heart failure No symptomatic ischemic heart disease Other: Not pregnant or nursing Fertile patients must use effective contraception HIV negative No uncontrolled infection No poorly controlled diseases (e.g., diabetes, systemic lupus erythematosus) No history of psychiatric disorders No other malignancies within the past 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix No concurrent severe medical problems No history of allergic reaction to topotecan and its derivatives

PRIOR CONCURRENT THERAPY: Biologic therapy: No other concurrent immunotherapy Chemotherapy: No prior topotecan At least 4 weeks since prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No other investigational drugs within 30 days of study No other concurrent investigational therapy except for basal cell skin cancer

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-02; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel C. Besa, MD, Study Chair — Drexel University College of Medicine
Locations (2):
- United States (2):
  - Medical College of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Medical College of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Besa E, Maiale C, Liman D, et al.: Early data on a new combination chemotherapy using topotecan, fludarabine, ARA-C and G-CSF for aggressive myelodysplastic syndromes in the elderly. [Abstract] Leuk Res 23 (Suppl 1): A-191, S72, 1999.